CLINICAL TRIAL: NCT04743791
Title: A Randomized, Placebo-controlled, Parallel Group Study Designed to Assess the Change in Mucociliary Clearance After 12 Weeks of Treatment With Dupilumab in Patients With Moderate to Severe Asthma
Brief Title: Measuring the Effect of Dupilumab Treatment on Mucociliary Clearance (MCC) in Subjects With Moderate to Severe Asthma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sally E. Wenzel MD (Other)
Responsible Party: Sponsor-Investigator, Sally E. Wenzel MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20020131
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dupilumab and placebo will be provided in identically matched 1.14 mL pre-filled syringes. To protect the blind, each treatment kit of 1.14 mL (dupilumab / placebo) glass pre-filled syringes will be prepared such that the treatments (dupilumab and its matching placebo) are identical and indistinguishable and will be labeled with a treatment kit number. The randomized treatment kit number list will be generated by Sanofi Regeneron
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Active Comparator): Two injections of Dupilumab will be administered at Week 0/Visit 3 as a loading dose. Subsequently one injection of Dupilumab will be given every 2 weeks ± 3 days at home by the patient. The doses of investigational product must be separated by ≥11 days to avoid an overdose.
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Two injections of placebo will be administered at Week 0/Visit 3 as a loading dose. Subsequently one injection of placebo will be given every 2 weeks ± 3 days at home by the patient. The doses must be separated by ≥11 day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab is supplied as a sterile aqueous solution for SC injection at the concentration of 175 mg/mL in glass pre-filled syringe to deliver 200 mg in 1.14mL.
  Arms: Dupilumab
Other: Placebo — Sterile placebo for dupilumab will be provided in identically matched glass pre-filled syringe to deliver 200 mg in 1.14mL, which will match dupilumab 200 mg (1.14mL).
  Other Names: Sucrose
  Arms: Placebo

SUMMARY:
Single center, randomized, placebo- controlled study to assess change in mucociliary clearance of moderate to severe asthma patients after treatment with dupilumab or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Moderate - Severe Th2 (Type 2) High asthma, as defined by Forced Expiratory Volume in one second (FEV1) <90% predicted, on medium to high dose inhaled corticosteroids (ICS) with or without a second controller
* Age > 18
* Inhaled steroid doses of 500micrograms (mcg) per day or more (Fluticasone equivalent)
* Reversibility >/= 12% at screening or within the past 2 years, or a positive methacholine challenge test within the past 2 years, or a positive methacholine challenge during screening
* FEV1/Forced Vital Capacity (FVC)<75%
* Blood Eosinophils (EOS) >300 cells per mm3
* Exhaled Nitric Oxide (FeNO) >25 parts per billion (ppb)
* Asthma Control Test (ACT) score <20

Exclusion Criteria:

* Pregnant, nursing, or unwilling to test for pregnancy
* Current smoker or >10 pack year smoking history
* Body Mass Index (BMI)>37
* Respiratory infection in the last 30 days
* Use of antibiotics or oral prednisone in the last 30 days
* Current or previous use of dupilumab
* Current or recent use of anti-IL-5 therapies
* Any other criteria that place the subject at unnecessary risk
* Diagnosis of other lung diseases including Chronic Obstructive Pulmonary Disease (COPD)
* History of non-skin cell cancer in the last 5 years
* Drug or alcohol addiction in the last 5 years
* Any other uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in mucociliary clearance (MCC) rate | Measured at 12 weeks after the start of treatment
  MCC is measured using an aerosol-based nuclear imaging technique

SECONDARY OUTCOMES:
Change in FEV1% predicted | Measured from baseline to 12 weeks after start of treatment
  Assessed using spirometry after bronchodilator administration.
Change in ACT score | Measured from baseline to 12 weeks after start of treatment
  Measured via the Asthma Control Test questionnaire. Scores range from 5 (poor control of asthma) to 25 (complete control of asthma).
Change in sputum eosinophils and T2 gene mean | Measured from baseline to 12 weeks after start of treatment
  Measured via sputum induction to obtain airway cells and fluid from patients.
Change in mucus plugging score by CT | Measured from baseline to 12 weeks after start of treatment
  Radiologists will visually assess the presence or absence of mucus plugging in segmental airways and will provide a mucus plugging score
Whole lung MCC90, AAC90 | Measured from baseline to 12 weeks after start of treatment
  Measured via mucociliary clearance imaging
Peripheral and central lung MCC90, MCC240, AAC90 | Measured from baseline to 12 weeks after start of treatment
  Measured via mucociliary clearance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Pittsburgh Asthma Institute at UPMC, Pittsburgh, Pennsylvania, United States